CLINICAL TRIAL: NCT02166814
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Combination of Fimasartan/Rosuvastatin in Comparison to Each Component Administered Alone in Patients With Essential Hypertension and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FRC-CT-301
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2014-06

CONDITIONS: Essential Hypertension, Dyslipidemia
MeSH Terms: conditions — Essential Hypertension; Dyslipidemias | interventions — fimasartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Fimasartan and Rosuvastatin (Experimental): Combination of Fimasartan and Rosuvastatin
  Interventions: Drug: Fimasartan and Rosuvastatin
- Fimasartan (Active Comparator): Fimasartan monotherapy
  Interventions: Drug: Fimasartan
- Rosuvastatin (Active Comparator): Rosuvastatin monotherapy
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan and Rosuvastatin
  Arms: Fimasartan and Rosuvastatin
Drug: Fimasartan
  Arms: Fimasartan
Drug: Rosuvastatin
  Arms: Rosuvastatin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combination of Fimasartan/Rosuvastatin in comparison to each component administered alone in patients with essential hypertension and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily signed informed consent for participating in this clinical trial
2. Male and female between 20 and 75 years old
3. Patients must have been confirmed essential hypertension and dyslipidemia at Screening visit (Visit1)
4. Patients who meet the following criteria of fasting LDL-C and blood pressure at Baseline visit (Visit3) assessment after undergoing the therapeutic lifestyle change.

   * Low risk group: the case that does not have any other risk factor apart from hypertension / LDL-C (mg/dL): ≥160, ≤250, Mean SiSBP(mmHg): ≥140, <180
   * Moderate risk group: the case that has more than or equal to one risk factor apart from hypertension and has the 10-year risk of less than 10% / LDL-C (mg/dL): ≥160, ≤250, Mean SiSBP(mmHg): ≥140, <180
   * Moderate high risk group: the case that has more than or equal to one risk factor apart from hypertension and has the 10-year risk between 10% and 20% / LDL-C (mg/dL): ≥130, ≤250, Mean SiSBP(mmHg): ≥140, <180
   * High risk group: the case of CHD (Coronary heart disease) or CHD risk equivalents

     * Risk factors include cigarette smoking, hypertension (BP≥140/90 mmHg or on antihypertensive medication), low HDL cholesterol (<40mg/dL), family history of premature CHD(CHD in male first-degree relative <55 years of age; CHD in female first-degree relative < 65 years of age), and age (men≥45 years; women ≥55 years). in case of HDL-C ≥60mg/dL, reduce 1 from the total number of risk factors.
     * Electronic 10 year risk calculators are available at www.nhlbi.nih.gov/guidelines/cholesterol
     * CHD includes history of myocardial infarction, unstable angina, coronary artery procedures (angioplasty or bypass surgery), or evidence of clinically significant myocardial ischemia.
     * CHD risk equivalents include atherosclerotic disease (peripheral arterial disease, abdominal aortic aneurysm and carotid artery disease [transient ischemic attacks or stroke of carotid origin or >50% obstruction of a carotid artery]), diabetes and 2+ risk factors with 10 year risk of over 20%
5. Subject must be able to understand the trial procedures and be willing to cooperate and complete the trial.

Exclusion Criteria:

1. Severe hypertension patients with mean siSBP ≥ 180mmHg and/or SiDBP ≥110mmHg at the assessment of Screening visit (Visit1) and/or Baseline visit (Visit3). Or patients with postural hypotension with manifestation.
2. Patients with the mean SiSBP from 3 times of measurement of over 20mmHg.
3. Secondary hypertension patients, but not limited to the following disease (example: renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc)
4. Secondary dyslipidemia: nephrotic syndrome, dysproteinemia, obstructive hepatopathy or Cushing's syndrome.
5. Patients with fasting TG ≥ 400mg/dL at Pre-Baseline visit (Visit2) assessment
6. History of myopathy, rhabdomyolysis or/and CK ≥ 2 times upper normal limit.
7. Use of lipid modifying drug within 4 weeks prior to Pre-Baseline visit (Visit2) and/or antihypertensive drug within 2 weeks prior to Pre-Baseline visit(Visit2)
8. Clinically significant renal function abnormality in the laboratory results at Pre-Baseline visit (i.e. serum creatinine ≥ 1.5 times upper normal limit), liver function abnormality (ALT, AST ≥ 2 times upper normal limit), severe fatty liver disease that requires medication.
9. Clinically significant hypokalemia(less than 3.5 mmol/L) or hyperkalemia (exceeded 5.5 mmol/L) measured at Pre-Baseline visit (Visit2)
10. Subjects with following surgical and internal disease that may affect absorption, distribution, metabolism or excretion of drugs and have conditions which include the following (but are not limited to): history of major gastrointestinal surgeries including gastrectomy, gastro-enterostomy or bowel resection, gastrointestinal bypass graft and stabling; current active gastritis, ulcer, gastrointestinal and rectal bleeding, presence of active inflammatory bowel syndrome or biliary obstruction with the past 12 months.
11. Subjects with depletion of body fluid or sodium ion not able to correct
12. Subjects with sever insulin-dependent Diabetes Mellitus(DM) or Chronic DM (HbA1c > 9% at Pre-Baseline visit, dosage of an oral hypoglycemic agent was modified within 12 weeks prior to screening visit , or currently use of active insulin treatment) or with hypothyroidism not able to correct.( TSH ≥ 1.5 times upper normal limit)
13. Subjects with severe heart disease (Heart failure New York Heart Association(NYHA) class 3 and 4), or history of any of the followings within the past 6 months; ischemic heart disease (e.g. angina pectoris, myocardial infarction), peripheral vascular disease, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft.
14. Subjects with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or any other clinical significant arrhythmia conditions at discretion of investigator
15. Subjects with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve stenosis, or mitral valve stenosis.
16. Subjects with severe cerebrovascular disorder (e.g. stroke, cerebral infarction or cerebral hemorrhage within the past 6 months)
17. Subjects with chronic inflammatory disease requiring an chronic anti-inflammatory therapy, past or current medical history with wasting disease, autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus) or connective tissue disease.
18. Subjects with known moderate or malignant retinosis (e.g. retinal hemorrhage, visual disturbance or retinal microaneurysm in the past 6 months)
19. Subjects with hepatitis B (including positive test for HBsAg), hepatitis C-positive
20. Subjects with history or evidence of abusing drugs or alcohol within the past 2 years.
21. Medical history with hypersensitivity to angiotensin II antagonist based drugs or HMG-CoA reductase inhibitor based drugs or any ingredient contained in these 2 drugs.
22. Medical history with clinically significant hypersensitivity to any components or other drugs on the investigational product or additives (yellow 5)
23. Subjects with hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
24. Pregnant women and lactating female.
25. Subjects planning pregnancy or childbearing potential who are not using effective contraceptive methods (surgical sterilized, intrauterine (contraceptive) device/condom or the combination of diaphragm and spermicidal agents)
26. Subjects who are participating in another trial or took other investigational product within 12 weeks prior to Screening visit
27. Medical history of all kinds of malignant tumor including leukemia and lymphoma in the past 5 years
28. A subject with other reasons not specified above that, ineligible to participate in this clinical trial at discretion of study investigators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change rate of LDL-C at week 8 of Fimasartan/Rosuvastatin combination administration from the Baseline to compare the one of Fimasartan 120mg single administration | 8 weeks from Baseline Visit
Change of SiSBP at week 8 of Fimasartan/Rosuvastatin combination administration from the Baseline to compare the one of Rosuvastatin 20mg single administration | 8 weeks from Baseline Visit

CONTACTS AND LOCATIONS:
Overall Officials: Dongjoo Oh, Study Chair — Korea University Guro Hospital
Locations (26):
- South Korea (26):
  - Seoul university Bundang hospital, Bundang
  - Dong-A university hospital, Busan
  - Inje Heaundai Paik hospital, Busan
  - Inje university Busan Paik hospital, Busan
  - The Catholic university of Korea Daegu hospital, Daegu
  - DongGuk university Gyeongju hospital, Gyeongju
  - DongGuk university Ilsan hospital, Ilsan
  - Inje university Ilsan Paik hospital, Ilsan
  - Gachon university Gil medical center, Incheon
  - Inha university hospital, Incheon
  - Jeju national university hospital, Jeju City
  - JeonNam university hospital, JeonNam
  - ChungNam university hospital, Jungnam
  - DanGuk university hospital, Jungnam
  - Kyungbook National university hospital, Kyungbook
  - Gangnam Severance hospital, Seoul
  - Jeil hospital, Seoul
  - Korea university Anam hospital, Seoul
  - Korea university Guro hospital, Seoul
  - Kyunghee university hospital, Seoul
  - Samsung Seoul hospital, Seoul
  - Seoul national university hospital, Seoul
  - Severance hospital, Seoul
  - The Catholic university St. Mary hospital, Seoul
  - Aju university hospital, Suwon
  - YoungNam university hospital, YoungNam

REFERENCES:
- [Derived] Rhee MY, Ahn T, Chang K, Chae SC, Yang TH, Shim WJ, Kang TS, Ryu JK, Nah DY, Park TH, Chae IH, Park SW, Lee HY, Tahk SJ, Yoon YW, Shim CY, Shin DG, Seo HS, Lee SY, Kim DI, Kwan J, Joo SJ, Jeong MH, Jeong JO, Sung KC, Kim SY, Kim SH, Chun KJ, Oh DJ. The efficacy and safety of co-administration of fimasartan and rosuvastatin to patients with hypertension and dyslipidemia. BMC Pharmacol Toxicol. 2017 Jan 5;18(1):2. doi: 10.1186/s40360-016-0112-7. PMID 28057081